CLINICAL TRIAL: NCT02936921
Title: Lyon Clinical Research Program on Maternal and Congenital Toxoplasmosis Based on the Toxo-Ly Cohort: Risks and Clinical Consequences, Prevention, Diagnosis and Treatment
Brief Title: Lyon Cohort of Maternal and Congenital Toxoplasma Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0569
Record Dates: First submitted 2016-09-06; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-09

CONDITIONS: Toxoplasmosis, Congenital
Keywords: Toxoplasma gondii; Toxoplasmosis; congenital; prenatal; screening; treatment; diagnosis
MeSH Terms: conditions — Toxoplasmosis, Congenital; Toxoplasmosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples with and without DNA are analyzed. blood samples taken during pregnancy to confirm maternal infection amniotic fluid analysed with PCR and inoculation to mice blood samples taken after birth for children born from a mother included in the cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pergravidic maternal infections: proven maternal infections: true seroconversions of profiles of recent infections
- Subjects free of congenital infection: children who whom all tests performed before birth, at birth and after birth confirmed the absence of congenital toxoplasmosis.
- Congenitally infected subjects: children for whom at least one test performed before birth, at birth or after birth demonstrated a congenital infection.

SUMMARY:
Several decades ago, France has made the choice to implement a national prevention program for congenital toxoplasmosis. The identification in their first trimester of pregnancy of all pregnant women who are susceptible to Toxoplasma infection has been mandatory since 1985. In 1992, the decision was made to extent the program to the monthly retesting of all women identified as not immune, in an attempt to reduce the number of severely infected children.

The systematic detection of all maternal and congenital infections has generated many questions from clinicians, biologists, parents and older patients, on the short and long-term prognosis of congenital toxoplasmosis, on the best tests to use to diagnose infections in mothers and children, on the efficacy of existing treatments, and on how to manage patients in the long-term.

The need to answer these many questions has prompted the medical team working within the laboratory and the outpatient department of the Parasitology Department at the Croix-Rousse Hospital in Lyon to implement a clinical research program. It is based on the systematic inclusion in our cohort of all pregnant women whose infection is confirmed, on their follow up, in order to monitor the outcome of pregnancy 2) and on the follow up of their children in order to confirm their infection or to rule it out. All congenitally infected subjects undergo clinical examinations, serological tests and ocular examination at least once a year without age limit.

The following data are prospectively collected in a dedicated database: gestational age at maternal infection and corresponding serological profile; type and dates of maternal treatment; findings of ultrasound tests and amniotic fluid analysis; serological and clinical findings at birth; types and dates of postnatal treatment; postnatal serological profiles; infection status at one year of age; long term clinical (ophthalmologic) et serological findings.

These data have allowed producing original findings on the risk of maternal-foetal transmission according to gestational age at maternal infection, on the long term ophthalmological outcome of congenital toxoplasmosis and to offer guidelines for the diagnosis, treatment and follow-up of maternal and congenital infections.

These efforts are still to be maintained in the future in order

* to further analyse the impact of puberty, pregnancy, or adult co-morbidities on the risk of ophthalmological events
* to increase precision around our risk estimates for materno-foetal transmission,
* to continue innovating in terms of diagnostic strategy to improve tests performances and reduce costs
* to explore new potential clinical outcomes such as neuropsychiatric disorders associated with congenital and postnatal infection
* to determine if infections due to oocysts could have different clinical outcomes than those due to the ingestion of cysts
* to assess the efficacy of treatments for maternal and congenital infections

ELIGIBILITY:
Inclusion Criteria:

* Confirmation in our laboratory of a maternal infection estimated to have occurred during pregnancy or during the 12 weeks preceding conception.

Exclusion Criteria:

* maternal :infection that could not be confirmed in our reference laboratory

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Systematic inclusion of all cases of pergravidic Toxoplasma infections identified through the French monthly retesting program and confirmed in our reference center.
  Systematic follow up of the outcome of pregnancy and systematic clinical and biological follow up of live born children, until the age of one year at least (to rule congenital toxoplasmosis in or out) or without limit for those who are recognized to have a congenital toxoplasmosis.
Sampling Method: Non-Probability Sample
Enrollment: 4030 (Estimated)
Dates: Start 1988-01; Primary Completion 2016-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Long term ophthalmological outcome of congenital infection | up to 37 years
  eye examinations are prospectively performed to detect lesions of retinochoroiditis or additional ocular lesions every three to six months in younger children and at least annually afterwards.
  A standardized form is used to report findings. Clinical examinations are performed at the same frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix Rousse Hospital, Lyon, France

REFERENCES:
- See also: Related Info — http://grossesse-toxoplasmose.univ-lyon1.fr/